CLINICAL TRIAL: NCT06542224
Title: Identifying Local Field Potential Biomarkers for Obsessive-compulsive Disorder Treatment With Deep Brain Stimulation
Acronym: DBS OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Botao Xiong, Assistant research fellow, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS-OCD-01
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; DBS; LFP; Biomarker
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- deep brain stimulation (Experimental)
  Interventions: Procedure: Deep Brain stimulation

INTERVENTIONS:
Procedure: Deep Brain stimulation — All subjects will receive bilateral surgical implantation of DBS system.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a complex and severe mental illness characterized by multiple symptoms and is considered a leading cause of non-fatal health loss. However, nearly 20% of patients do not respond to standard pharmacological or psychological treatments. Currently, we lack objective brain-based biomarkers. To address this issue, we used a novel device for electrophysiology recording and applied deep brain stimulation (DBS) to 16 OCD patients. In this study, we aim to use long-term invasive neural signal collection and machine learning techniques to reveal the complex relationship between these signals and OCD symptoms. By applying advanced machine learning algorithms, our goal is to establish highly accurate prediction models to identify biomarkers associated with the occurrence and progression of OCD. The research will focus on the spatiotemporal features of neural signals and build personalized OCD decoding models based on individual differences through the integration and analysis of large-scale data. By delving into the information contained in neural signals, we hope to provide academic and practical innovations for the development of personalized treatment approaches for OCD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with OCD according to the criteria in the DSM-5.
2. Age between 18 and 65 years.
3. Duration of illness of more than 3 years.
4. Ineffectiveness of systematic treatment with three types of serotonin reuptake inhibitors (including clomipramine) and augmentation agents, with no improvement after continuous high-dose serotonin reuptake inhibitor treatment for more than 12 weeks, or the occurrence of severe adverse drug reactions during treatment.
5. Ineffectiveness of CBT treatment or repeated refusal of CBT treatment.
6. Y-BOCS total score of 25 or higher.
7. Significant impairment in social functioning, such as inability to work or attend school, or a noticeable decline in personal life skills.
8. No severe impairment in insight, and capable of signing informed consent and surgery consent forms.

Exclusion Criteria:

1. Presence of bipolar disorder, schizoaffective disorder, schizophrenia, or other psychotic disorders.
2. Severe personality disorders.
3. Severe physical illnesses or organic brain diseases.
4. Diagnosis of alcohol or substance abuse and dependence according to DSM-IV criteria within one year prior to screening.
5. Study participants with contraindications for surgery, such as major medical comorbidities or inability to discontinue anticoagulant medications.
6. Preoperative head MRI showing significant structural abnormalities.
7. Contraindications for MRI examination (excluding the DBS implant or stimulator itself).
8. Pregnancy or breastfeeding.
9. Study participants currently enrolled in another research study unrelated to the current study.
10. Any condition that currently or in the future might endanger the safety of the study participant or prevent the successful participation in the study (including family support, medical, psychological, social, or geographical factors).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-03 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Identifying an electrophysiological biomarker of OCD | 30 days
  Percentage of patients in which an electrophysiological biomarker of OCD can be identified before initial DBS

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - West CHina Hospital，Sichuan University, Chengdu, Sichuan
  - The First People's hospital of Longquanyi District, Chengdu, Sichuan
  - Zigong Fifth People's Hospital, Zigong, Sichuan
  - Zigong Fourth People's Hospital, Zigong, Sichuan